CLINICAL TRIAL: NCT06708026
Title: Evaluation of a Home-based Action Observation and Motor Imagery Intervention on Cognitive Function and Depression Among Adults with Spinal Cord Injury: a Pilot Randomized Controlled Trial
Brief Title: Evaluation of a Home-based AOMI Intervention on Cognitive Function and Depression Among Adults with SCI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSEARS20240716007-01; P0051299 (Other Grant/Funding Number: The Hong Kong Polytechnic University Fund)
Record Dates: First submitted 2024-11-19; First posted 2024-11-27 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2024-11

CONDITIONS: Spinal Cord Injuries (SCI); Depression; Motor Imagery; Cognitive Functions
MeSH Terms: conditions — Spinal Cord Injuries; Depression

STUDY DESIGN:
Intervention Model Description: We aim to have two study groups. Forty-six participants will be randomly assigned to either the intervention group, which will receive an 8-week AOMI intervention combined with basic wheelchair exercises, or the control group, which will watch landscape videos and perform basic wheelchair exercises. The intervention duration, number of sessions, and frequency of the control group are the same as the intervention group.
Who Masked: Outcomes Assessor
Masking Description: Participants and the researcher who will enroll in the intervention process and conduct the qualitative interview will not be blinded. The data analyst and the baseline and outcome assessor will be blinded from the group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): For each session, participants will be required to conduct a ten-minute basic wheelchair exercise followed by a twenty-minute AOMI training at home. The whole intervention will last for eight weeks, three times a week.
  Interventions: Behavioral: Action Observation and Motor Imagery (AOMI) training; Behavioral: Basic wheelchair exercises
- Control group (Active Comparator): For each session, participants will be required to conduct a ten-minute basic wheelchair exercise, followed by 20 minutes of watching landscape videos in their homes. The whole intervention will last for eight weeks, three times a week.
  Interventions: Behavioral: Basic wheelchair exercises; Behavioral: Watch landscape videos

INTERVENTIONS:
Behavioral: Action Observation and Motor Imagery (AOMI) training — Participants will watch home-based exercise videos and simultaneously imagine themselves performing these exercises in their minds by following verbal instructions in the videos, without actual execution.
  Arms: Intervention group
Behavioral: Basic wheelchair exercises — A set of low-intensity warm-up wheelchair exercises developed specifically for survivors with spinal cord injury
Behavioral: Watch landscape videos — A set of landscape videos
  Arms: Control group

SUMMARY:
The investigators propose a pilot randomized clinical trial to determine if adults with spinal cord injury (SCI) show improved cognitive function and depression following home-based Action Observation and Motor Imagery (AOMI) training. It is hypothesized that the home-based AOMI intervention will show satisfactory feasibility and acceptability. They also hypothesize that AOMI training can be used as a rehabilitative tool for improving cognitive function and depression in adults with SCI, because it engages and strengthens similar neural systems as actual exercise.

DETAILED DESCRIPTION:
This study is an assessor-blinded, two-arm pilot randomized controlled trial with repeated measures (pre-, post-intervention, and 1-month follow-up). This study aims to evaluate the preliminary effects of a home-based AOMI intervention on SCI adults' cognitive function and depression. Forty-six SCI adults will be randomized into the intervention group, receiving an 8-week AOMI intervention combined with basic wheelchair exercises, or the control group, receiving basic wheelchair exercises with the same duration, number of sessions, and frequency as the intervention group. One-on-one qualitative interviews will be implemented post-intervention to evaluate participants' feelings about the effectiveness of their cognitive function and emotional status, their views about opinions of the study's acceptability, strengths, limits, and recommendations for further improvement of the program. The primary outcomes of intervention effectiveness include cognitive function and depression; secondary outcomes include multi-model magnetic resonance imaging (MRI) acquisition, chronic pain, motor imagery ability, and self-efficacy for exercise.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of SCI according to the International Standards for the Neurological Classification of SCI with confirmation by computed tomography/magnetic resonance imaging;
* At least 18 years old;
* With stable spinal systems and good vital signs, and currently living in the community and having SCI for more than 6 months;
* No contraindications to undergoing MRI examination (e.g., no metal or electronic devices in the body, not pregnant, and absence of claustrophobia);
* Having a mobile Internet terminal (usually a smartphone) and proficient independent or caregiver-assisted usage;
* Able to communicate in Cantonese and to provide informed consent.

Exclusion Criteria:

* Having severe problems in hearing, verbal communication, or vision;
* Engaged in ongoing psychotherapy or any other physiotherapy/ exercise/ relaxation interventions;
* Physically active for more than 150 minutes moderate-intensity exercise per week;
* Diagnosis of mental disorders or substance misuse;
* With severe cognitive impairment (Hong Kong Montreal Cognitive Assessment (HK-MoCA) score ≤ 18.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | Pre-intervention
  The recruitment rate refers to the percentage of participants who give consent after determining their eligibility.
Retention rate | 1-month follow-up
  The retention rate will be determined by dividing the number of individuals who finish the research by the total number of participants who consent.
Dropout rate | 1-month follow-up
  The dropout rate will be determined by the number of individuals who withdraw post-randomization divided by the total number of participants who consented.
Number of participants with adverse events | During the intervention
  The count of participants who reported at least one adverse event related to the intervention, including severe dizziness, fatigue, and pain.
Intervention satisfaction | Immediately after intervention (an average of two months)
  The intervention satisfaction will be assessed using an 8-item Client Satisfaction Questionnaire employing a four-point Likert scale, alongside one-on-one qualitative interviews. The total possible score on the 8-item Client Satisfaction Questionnaire ranges from 8 to 32, with higher scores indicating greater levels of satisfaction.
Adherence rate | Immediately after intervention (an average of two months)
  The adherence rate refers to the percentage of participants completing a minimum of 60% of interventions, equivalent to at least 15 sessions.
Global cognitive function | Baseline, immediately after intervention (an average of two months), and 1-month follow-up
  The Chinese version of Neuropsychiatry Unit Cognitive Assessment Tool (NUCOG) will be used. This tool comprises 21 items in 5 cognitive domains: attention, visuoconstructional, memory, executive, and language. Scores for each of the domains range between 0 and 20, adding up to a total NUCOG score out of 100. Higher scores indicate higher levels of cognitive function.
Depression | Baseline, immediately after intervention (an average of two months), and 1-month follow-up
  The level of depression will be assessed by version 2 of the Beck Depression Inventory (BDI-II), which consists of 21 items assessing 2 factors (cognitive and affective, and somatic symptoms). The total possible score of BDI-II is 0 to 63; higher scores reflect higher levels of depression.

SECONDARY OUTCOMES:
The Digit Span Test [Forward Span] | Baseline, immediately after intervention (an average of two months), and 1-month follow-up
  The Digit Span Test [Forward Span] will be used to assess attention, concentration, and short-term memory. The examiner will pronounce a list of digits at a rate of approximately one digit per second, and subjects are required to immediately repeat the list in the same order. The Digit Span Test scores range from 0 to 9. The higher scores mean a better outcome.
The Digit Span Tests [Backward Span] | Baseline, immediately after intervention (an average of two months), and 1-month follow-up
  The backward digit span task measures visuospatial integration and working memory; hence, the backward digit span task is a more appropriate measure for executive function. The backward digit span task uses the same procedure as the Digit span forward task, except that in this case, subjects have to reproduce the sequence of digits in reverse order, and the longest list consists of nine items. The Digit Span Test scores range from 0 to 9.
The Stroop Color Word Test | Baseline, immediately after intervention (an average of two months), and 1-month follow-up
  The Stroop Color Word Test will be used to measure executive function and attention. It will be determined by subtracting the Color (congruent trials) from the Color-Word (incongruent trials) scores. It is a measure of response competition and interference. Scoring is based on the time it takes to read (complete) incongruent trials relative to congruent trials. A negative mean value reflects an improvement in performance after the intervention. A positive mean value reflects a decrease in performance after the intervention.
The oral version of the Symbol Digit Modalities Test | Baseline, immediately after intervention (an average of two months), and 1-month follow-up
  This test will be used to assess cognitive processing speed. The participant will be given 90 seconds to verbally match symbols with digits as quickly as possible. The correct verbal responses will be recorded. A larger number of correct answers given within the time limit represents better switching attention and information-processing speeds in an individual.
Change in gray matter cortical thickness | Baseline, immediately after intervention (an average of two months)
  Change in mean cortical thickness obtained from T1-weighted structural images. A positive mean value reflects an increase in cortical thickness post-intervention, and a negative mean value reflects a decrease in cortical thickness post-intervention.
Change in white matter integrity | Baseline, immediately after intervention (an average of two months)
  Change in white matter integrity obtained from diffusion-weighted imaging. Increased white matter integrity is associated with improved cognitive performance, whereas decreased white matter integrity is associated with decreased cognitive performance.
Change in white matter hyperintensities | Baseline, immediately after intervention (an average of two months)
  Change in white matter hyperintensities obtained from Fluid-Attenuated Inversion Recovery imaging. Increased white matter hyperintensities may be indicative of unfavorable outcomes.
Change in Blood-oxygen-level-dependent (BOLD) signal during Action Observation and Motor Imagery task conditions | Baseline, immediately after intervention (an average of two months)
  Change in blood-oxygen-level-dependent (BOLD) signal (neuroplasticity) during performing mental imagination of the action while watching the video will be measured using task-based functional magnetic resonance imaging (fMRI). The mean values reported are changes in factor scores that reflect the overall change in the BOLD signal pre- to post-intervention. Positive values reflect an increase in BOLD signal post-intervention, whereas negative mean values reflect a decrease in BOLD signal post-intervention. There are no minimum or maximum values, ranges, or thresholds associated with the BOLD measure.
Change in functional connectivity features or neural networks | Baseline, immediately after intervention (an average of two months)
  Change in functional connectivity features or neural networks will be measured using resting-stated fMRI.
Pain | Baseline, immediately after intervention (an average of two months), and 1-month follow-up
  The Chinese version of the Brief Pain Inventory (BPI-C) will be used to assess the pain severity and interference. The total scores for pain severity (4 items) and interference (7 items) are measured with a 11-point scale (from 0 = no pain/interference to 10 = worst pain/interference imaginable), where higher scores represent more violent pain.
Self-efficacy for exercise | Baseline, immediately after intervention (an average of two months), and 1-month follow-up
  The 9-item Chinese version of the self-efficacy for exercise will be used to evaluate participants' confidence level (from 0 not confident to 10 very confident) regarding engaging in regular exercise.
Motor imagery ability | Baseline, immediately after intervention (an average of two months), and 1-month follow-up
  The short version of the Kinesthetic and Visual Imagery Questionnaire (the KVIQ-10) will be used to evaluate the participants' motor imagery ability.

CONTACTS AND LOCATIONS:
Locations (1):
- School of Nursing, The Hong Kong Polytechnic University, Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hu Y, Li Y, Tao R, Hsu CL, Craig A, Lam CY, Kahraman T, Leung AYM. Effects and mechanisms of a home-based action observation and motor imagery intervention on cognitive function and depression in spinal cord injury: a pilot randomized controlled trial protocol. Front Neurol. 2025 May 16;16:1578323. doi: 10.3389/fneur.2025.1578323. eCollection 2025. PMID 40452762